CLINICAL TRIAL: NCT01829841
Title: A Randomized, Positive-controlled, Double-blind, Multicenter, Phase II Study of Famitinib as First/Second Line Treatment in Patients With Advanced Metastatic Renal Cell Cancer
Brief Title: A Study of Famitinib in Patients With Advanced Metastatic Renal Cell Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Collaborators: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FMTN-II-MRCC
Record Dates: First submitted 2013-04-08; First posted 2013-04-11 (Estimated); Last update posted 2018-05-03 (Actual); Status verified 2013-04

CONDITIONS: Renal Cell Cancer; Metastatic Renal Cell Cancer
Keywords: MRCC; Metastatic Renal Cell Cancer; Famitinib; Sunitinib
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — famitinib; Sunitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Famitinib (Experimental): Famitinib 25 mg qd p.o., 6 weeks per cycle.The treatment continued until disease progression or intolerable toxicity happened or patients withdrawal of consent.
  Interventions: Drug: Famitinib
- Sunitinib (Active Comparator): Sunitinib 50 mg qd p.o., 4 weeks out of 6.The treatment continued until disease progression or intolerable toxicity happened or patients withdrawal of consent.
  Interventions: Drug: Sunitinib

INTERVENTIONS:
Drug: Famitinib — Famitinib 25 mg p.o. qd
  Arms: Famitinib
Drug: Sunitinib — Sunitinib 50 mg p.o. qd
  Arms: Sunitinib

SUMMARY:
* Famitinib is a tyrosin-inhibitor agent targeting at c-Kit, VEGFR2, PDGFR, VEGFR3, Flt1 and Flt3. Phase I study has shown that the toxicity is manageable.
* The purpose of this study is to compare the efficacy and safety profile between Famitinib and Sunitinib in patients with metastatic renal cell carcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically confirmed advanced renal cell carcinoma including clear cell component and not available for surgery
* First-line therapy or second-line treatment (second-line treatment e.g chemotherapy or cytokine therapy as first-line treatment failure or resistant patients)
* With measurable disease (using RECIST1.0 standard conventional CT scan ≥ 20 mm, spiral CT scan ≥ 10mm, target lesion did not receive radiation therapy, cryotherapy)
* Male or female, age ≥18 and ≤75
* ECOG 0-1
* Life expectancy ≥ 3 months
* Subjects received surgery, chemotherapy, radiation therapy, cytokines treatment caused the damage has been restored, the time interval ≥ 4 weeks, and the wound has completely healed
* Normal major organ function
* Signed and dated informed consent

Exclusion Criteria:

* Previously received targeted therapy of the metastatic renal cell carcinoma (such as sunitinib, Sorafenib)
* Past or suffering from other cancer, but other than cure basal cell carcinoma and cervical carcinoma in situ
* Participated in other clinical trials within four weeks
* A variety of factors that affect the oral medication (such as inability to swallow, gastrointestinal resection, chronic diarrhea and intestinal obstruction)
* Known brain metastases, spinal cord compression, cancer, meningitis, or screening CT or MRI examination revealed brain or leptomeningeal disease
* Patients with hypertension (systolic blood pressure> 140 mmHg, diastolic blood pressure> 90 mmHg). Patients with more than Class I, myocardial ischemia or myocardial infarction, arrhythmia (including QT interval ≥ 440ms) and class I heart failure.
* Urine protein ≥ + + and confirmed the 24-hour urinary protein>1.0 g
* Coagulopathy with bleeding tendency (such as active peptic ulcer) or are receiving thrombolytic or anticoagulant therapy
* Previous hyperactivity / venous thromboembolic events, such as cerebrovascular accident (including transient ischemic attacks), deep vein thrombosis and pulmonary embolism
* The preexisting abnormal thyroid function, even in the case of medication still can not be maintained within the normal range
* With a history of abuse of psychotropic drugs or mental disorders
* Patients with Hepatitis B or Hepatitis C
* History of immunodeficiency, including HIV testing positive or suffering from acquired, congenital immunodeficiency disease, or a history of organ transplantation

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2011-05; Primary Completion 2013-04 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Objective Response Rate | 18 weeks

SECONDARY OUTCOMES:
Progress free survival (PFS) | 3 years
Disease Control Rate (DCR) | 3 years
Overall Survival (OS) | 3 years
Quality of Life | 42-day cycle visit until disease progress
Number of Participants with Adverse Events as a Measure of Safety | 3 years

OTHER OUTCOMES:
body vitals, laboratory parameters | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Jinwan Wang, M.D, Study Chair — Cancer Institute and Hospital, Chinese Academy of Medical Sciences; Jianhui Ma, M.D, Study Chair — Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Locations (1):
- Cancer Institute and Hospital Chinese Academy of Medical Sciences, Beijing, China